CLINICAL TRIAL: NCT02945930
Title: A Prospective Multicenter, Open Study on the Safety and Efficacy of "Compont Medical Glue" in the Treatment of Esophagogastric Varices
Brief Title: Study the Safety and Efficacy of "Compont Medical Glue" in the Treatment of Esophagogastric Varices
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Director of department of Gastroenterology, Shanghai Zhongshan Hospital
Other Study IDs: CSY-2016-ZZJ
Record Dates: First submitted 2016-10-11; First posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal and Gastric Varices
Keywords: Enbucrilate; Esophageal and Gastric Varices; Endoscopy; Safety; Efficacy
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To observe the Safety and Efficacy of Compont Medical Glue in the Treatment of Esophagogastric Varices.

DETAILED DESCRIPTION:
"Compont Medical Glue" is a kind of histoacryl producted by Compont Company. It has been used to treat esophagogastric varices for several years. This study is a prospective multicenter,open study on the safety and efficacy of Compont Medical Glue in the treatment of esophagogastric varices. Weather the patient receiving injection of Compont Medical Glue is according to the degree of esophageal-gastric varices and is decided by the experienced endoscopic physicians. No additional intervention will be given to the patients, no matter whether patients are participated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Esophagogastric varices caused by portal hypertension with or without history of bleeding and no matter whether emergency bleeding.
* Patients may need to receive injection of histoacryl.
* Have signed informed consent.

Exclusion Criteria:

* Allergic to formaldehyde or cyanoacrylate.
* Women who are pregnant or breast-feeding.
* With contraindications of endoscopic exam.
* Computed tomography(CT)/Computed tomography angiography(CTA) shows that patient with severe portosystemic shunt.
* Large amount of blood accumulated in the stomach severely affects the endoscopic vision clarity.
* Other reasons that researcher think the patient is unsuitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophagogastric varices caused by portal hypertension who might need to receive endoscopy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The Occurrence Rate Of Different Adverse Event | Up to 2 months after the injection of histoacryl.
  Chest Pain/Epigastric Pain: Appears within 24 hours after injection of Compont Medical Glue and painkillers are used.
  Short-term Haemorrhage: Appears within 24 hours after injection of Compont Medical Glue.
  Glue Injection Related Bleeding: Appears within 2 months after injection of Compont Medical Glue confirmed by endoscopy.
  Fever: Patient has a fever over 38.0℃ within 3 days after injection of Compont Medical Glue.
  Ectopic Embolization: Appears within 3 days after injection of Compont Medical Glue and was confirmed by auxiliary examinations.
  Local Mucosal Necrosis: Local mucosal necrosis or ulcer appears around the injection poin within 2 months after injection of Compont Medical Glue.

SECONDARY OUTCOMES:
Bleeding Rate | 14 days and 2 months after injection of histoacryl.
  Data are analyzed separately as 14 days and 2 months for those patients who received endoscopic therapy for primary prevention of gastroesophageal varices bleeding.
Rebleeding Rate | 14 days and 2 months after injection of histoacryl.
  Data are analyzed separately as 14 days and 2 months for those patients who received endoscopic therapy for secondary prevention of gastroesophageal varices bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Monsanto P, Almeida N, Rosa A, Macoas F, Lerias C, Portela F, Amaro P, Ferreira M, Gouveia H, Sofia C. Endoscopic treatment of bleeding gastric varices with histoacryl (N-butyl-2-cyanoacrylate): a South European single center experience. Indian J Gastroenterol. 2013 Jul;32(4):227-31. doi: 10.1007/s12664-012-0191-3. Epub 2012 Jul 6. PMID 22766643
- [Background] Jun CH, Kim KR, Yoon JH, Koh HR, Choi WS, Cho KM, Lim SU, Park CH, Joo YE, Kim HS, Choi SK, Rew JS. Clinical outcomes of gastric variceal obliteration using N-butyl-2-cyanoacrylate in patients with acute gastric variceal hemorrhage. Korean J Intern Med. 2014 Jul;29(4):437-44. doi: 10.3904/kjim.2014.29.4.437. Epub 2014 Jun 27. PMID 25045291
- [Background] Khawaja A, Sonawalla AA, Somani SF, Abid S. Management of bleeding gastric varices: a single session of histoacryl injection may be sufficient. Eur J Gastroenterol Hepatol. 2014 Jun;26(6):661-7. doi: 10.1097/MEG.0000000000000080. PMID 24732750